CLINICAL TRIAL: NCT07007416
Title: Impact of Supraphysiological Estradiol Levels on Cardiac Electrophysiological Parameters During IVF: A Prospective Observational Study
Brief Title: Impact of Supraphysiological Estradiol on ECG in IVF Patients
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Dilay Gök Korucu, Assistant Prof. of Obstetrics and Gynecology, Konya City Hospital
Other Study IDs: 2024/026
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: In Vitro Fertilization; Estradiol; Cardiac Electrophysiology; Electrocardiography (ECG); Reproductive Endocrinology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aimed to evaluate the effects of supraphysiological estradiol (E2) levels, induced by gonadotropin therapy during IVF, on cardiac electrophysiological parameters. Sixty-two women aged 18-40 undergoing IVF treatment at Konya City Hospital between December 2024 and January 2025 were included.

ECG recordings were performed twice: once before gonadotropin stimulation and again on the day of hCG administration, when peak E2 levels were expected. Routine blood tests and hormone levels were also evaluated. Patients with obesity, cardiovascular disease, chronic illness, or medication use were excluded.

After treatment, significant increases were observed in PR interval, J-Tpeak, QTc, and Tp-e values. E2 changes showed a moderate negative correlation with QTc and a low positive correlation with J-Tpeak.

The results suggest that elevated E2 levels during IVF may affect cardiac electrophysiology, highlighting the need for careful monitoring in women with cardiac risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 40 years

Undergoing IVF treatment at Konya City Hospital between December 2024 and January 2025

No cardiac pathology based on cardiology consultation

Eligible for controlled ovarian stimulation using a short antagonist protocol

Provided informed consent

Exclusion Criteria:

- Age under 18 or over 40 years

Baseline estradiol level > 50 ng/L on day 2 of menstrual cycle

Presence of any known chronic diseases (e.g., diabetes mellitus, hypertension, rheumatologic disorders, thyroid disorders)

Use of any medications other than those used for IVF

Current smoker or alcohol user

Family history of cardiac disease or sudden cardiac death

Personal history of myocardial infarction, angina, heart failure, or any structural heart disease

History of cardiac surgery or coronary intervention

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged 18 to 40 years undergoing in vitro fertilization (IVF) treatment at the IVF Unit of Konya City Hospital. All participants were free of known cardiovascular or chronic systemic diseases and met the inclusion criteria for controlled ovarian stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in QTc Interval Before and After Gonadotropin-Induced Estradiol Elevation | Approximately 8-12 days from baseline to post-treatment ECG
  QTc interval will be measured via 12-lead electrocardiography (ECG) at two timepoints: (1) on menstrual cycle day 2-3 prior to gonadotropin stimulation (baseline), and (2) on the day of hCG administration when estradiol reaches peak levels. The difference between pre- and post-treatment QTc values will be calculated.

SECONDARY OUTCOMES:
Change in PR Interval Following Gonadotropin-Induced Estradiol Elevation | Approximately 8-12 days
  PR interval will be assessed using standard 12-lead ECG both before and after gonadotropin stimulation. Measurements will be taken on menstrual day 2-3 and again on the day of hCG administration to evaluate PR interval prolongation in response to elevated estradiol levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dilay Gök Korucu, M.D., Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No